CLINICAL TRIAL: NCT06449170
Title: BIAMEX: Discovery of Biomarkers of Intake of Highly Consumed Foods in Mexico by Untargeted Metabolomics
Brief Title: Discovery of Biomarkers of Intake of of Highly Consumed Foods in Mexico
Acronym: BIAMEX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Natalia Vázquez Manjarrez, Researcher in Medical Sciences, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 4044
Record Dates: First submitted 2024-05-22; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Nutrition, Healthy; Diet Habit; Diet, Healthy; Dietary Exposure
Keywords: metabolomics; nutrition; dietary biomarkers; dietary exposure
MeSH Terms: conditions — Feeding Behavior | interventions — Amaranth Dye

STUDY DESIGN:
Intervention Model Description: This is a randomized, open, crossover, and controlled design study. A total of 12 healthy subjects (six males and six females) aged 18-40 years with a BMI of 18.5-24.9 kg/m^2 were recruited. Participants underwent seven interventions (each featuring one of the selected foods or a control beverage), with a washout period of 7 days between interventions.
  Each intervention is as follows:
  150g of mango + 150ml of control beverage, 120g of avocado + 150ml of control beverage, 300g of cooked nopal + 150ml of control beverage, 3 corn tortillas + 150ml of control beverage, 3 guavas + 150ml of control beverage,
  ½ cup of amaranth + 150ml of control beverage, 290ml of control beverage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Mango Ataulfo (Other): 150g of mango Ataulfo plus 150 ml of control beverage (Supportan® Drink Cappuccino) plus 15ml of sunflower seed oil
  Interventions: Other: Mango Ataulfo
- Avocado Hass (Other): 120g of avocado hass plus 150ml of control beverage (Supportan® Drink Cappuccino)
  Interventions: Other: Avocado Hass
- Boiled Nopal (Other): 300g of boiled nopal plus 150 ml of control beverage (Supportan® Drink Cappuccino) plus 18ml of sunflower seed oil
  Interventions: Other: Nopal
- Corn Tortilla (Other): 3 pieces of corn tortilla plus 150 ml of control beverage (Supportan® Drink Cappuccino) plus 2ml of sunflower seed oil
  Interventions: Other: 3 corn tortilla
- Guava (Other): 3 pieces of guava plus 150 ml of control beverage (Supportan® Drink Cappuccino) plus 16ml of sunflower seed oil
  Interventions: Other: Guava
- Amaranth (Other): 1/2 cup of amaranth plus 150 ml of control beverage (Supportan® Drink Cappuccino) plus 35ml of sunflower seed oil
  Interventions: Other: Amaranth
- Supportan® DKN Cappuccino (Other): 290ml of control beverage (Supportan® Drink Cappuccino)
  Interventions: Dietary Supplement: Control Beverage (Supportan Drink ® Capuccino)

INTERVENTIONS:
Other: Mango Ataulfo — In this intervention, subjects consumed 150g of mango Ataulfo plus 150 ml of control beverage (Supportan® Drink Cappuccino). The addition of the control beverage has the purpose of providing energy intake and limiting the noise that the control beverage may contribute to the metabolomic profile in urine and serum.
  Arms: Mango Ataulfo
Other: Avocado Hass — In this intervention, subjects consumed 120g of avocado hass plus 150 ml of a control beverage (Supportan® Drink Cappuccino). The addition of the control beverage provides energy intake and limits the noise that the beverage may contribute to the metabolomic profile in urine and serum.
  Arms: Avocado Hass
Other: Nopal — In this intervention, subjects consumed 300g of cooked nopal and 150 ml of control beverage (Supportan® Drink Cappuccino). The addition of the control beverage provides energy intake and limits the noise that the beverage may contribute to the metabolic profile in urine and serum.
  Arms: Boiled Nopal
Other: 3 corn tortilla — In this intervention, subjects consumed 3 corn tortillas and 150 ml of control beverage (Supportan® Drink Cappuccino). The addition of the control beverage provides energy intake and limits the noise that the beverage may contribute to the metabolic profile in urine and serum.
  Arms: Corn Tortilla
Other: Guava — In this intervention, subjects consumed 3 guavas and 150 ml of control beverage (Supportan® Drink Cappuccino). The addition of the control beverage provides energy intake and limits the noise that the beverage may contribute to the metabolic profile in urine and serum.
  Arms: Guava
Other: Amaranth — In this intervention, subjects consumed 1/2 cup of amaranth and 150 ml of control beverage (Supportan® Drink Cappuccino). The addition of the control beverage provides energy intake and limits the noise that the beverage may contribute to the metabolic profile in urine and serum.
  Arms: Amaranth
Dietary Supplement: Control Beverage (Supportan Drink ® Capuccino) — In this intervention, subjects consumed 290ml of Supportan Drink ® Capuccino to act as a control for the metabolomic profiling in urine and serum.
  Arms: Supportan® DKN Cappuccino

SUMMARY:
To determine diet-health associations, researchers rely on information obtained from dietary instruments, such as the 24-hour recall (R24H), food frequency questionnaires (FFQ) and food diaries, in clinical studies. However, it is widely recognized that the information provided by the different instruments is biased by different factors including recall errors and respondent burden. The impact of the variability produced by this bias decreases the robustness of diet-health associations which results in the creation of less efficient standards and recommendations for our population. To address this, the discovery of biomarkers of food intake (BFIs) is an objective tool that indicates exposure to specific foods or various dietary patterns. BFIs allow the calibration of dietary information to obtain the real consumption of the individual and thus clarify the relationship between different pathologies of interest and the intake of different foods. BIAMEX will initially focus on the discovery of BFIs of nopal, corn tortilla, mango, avocado, guava and amaranth. For this purpose, a controlled crossover intervention study is being carried out with the 6 foods to be investigated where 24h urine and plasma samples are being collected. Subsequently, the samples collected will be analyzed by mass spectrometry.

DETAILED DESCRIPTION:
The BIAMEX study aims to address the challenge of improving the accuracy of dietary assessment, a critical factor in misunderstanding the relationship between diet and disease. Traditional dietary assessment tools, such as 24-hour recalls and food frequency questionnaires, are susceptible to biases related to their retrospective nature, such as memory errors and respondent burden. To overcome these limitations, BIAMEX focuses on discovering biomarkers on food intake (BFIs) for foods that originate in our country and are highly consumed by the population. This project will investigate the BFIs for nopal, corn tortilla, mango, avocado, guava, and amaranth.

This exploratory study employs a randomized, open, crossover, controlled design to investigate the metabolomic changes in urine and serum samples from healthy volunteers following the consumption of the selected foods. The interventions aim to assess the impact of each food intake on the metabolomic profile of the participants using an untargeted approach with liquid chromatography-mass spectrometry.

Participants were briefed at the Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán" on the study's aims, procedures, and benefits before providing informed consent. Subsequent steps included clinical history documentation and blood sampling for eligibility assessment, focusing on fasting glucose, cholesterol levels, and other health indicators. Volunteers underwent seven distinct food interventions in a randomized manner, including mango, avocado, nopal, corn tortillas, guavas, amaranth, and Supportan® drink Cappuccino as the control. This beverage was chosen to avoid metabolomic overlap with the different foods, ensuring distinct biomarker detection. Preceding the intervention days, subjects followed a low-polyphenol diet, excluding test foods and phytochemicals-rich items such as tea, coffee, or chocolate, culminating in a standardized dinner. On the intervention day, subjects arrived fasting at the institution and provided a baseline serum and urine samples. Then, subjects were provided with the test food, after which urine and serum samples were collected at 1h, 2h,4h, 6h postprandially on site. After the six-hour timepoint, the catheter was removed, and a standardized lunch was provided. Subjects continued to collect urine samples at home, corresponding to the 12h and 24h urine collection, using materials provided by the investigation team. Additionally, subjects received dietary instructions and menus to follow for the rest of the day. On the day after the intervention, subjects returned to the institution to deliver the urine collections and to provide the last serum sample corresponding to the 24-hour timepoint. Once the sample was collected, subjects were provided with a complimentary breakfast, and their habitual diet was resumed. This experimental procedure was repeated for each food separated by a 7-day wash-out period.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy males and females
* BMI >18.5 and < 25 kg/m2
* Willing/able to consume all test foods and the standardized meals

Exclusion Criteria:

* Smokers
* Diagnosed health condition (chronic or infectious disease)
* Taking nutritional supplements (e.g. vitamins, minerals) several times a week.
* Taking medication.
* Pregnant, lactating.
* Antibiotics treatment within 3 months prior to intervention.
* Vegetarians, as standardized meals will contain meat.
* Not willing to follow nutritional restrictions, including drinking alcohol during study days
* Allergic to foods of interest

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic profiling of urine samples after intake of mango, amaranth, nopal, corn tortilla, avocado, and guava, detected as mass-to-charge signals (cps) by an untargeted metabolomics approach over 24 hours post-intake. | Before intake of foods 00 hours to 24 hours after intake.
  Given the absence of a priori knowledge of specific urinary biomarkers of intake for mango, nopal, amaranth, avocado, corn tortilla, and guava, an untargeted metabolomics approach will be employed to identify them. As an exploratory approach, this methodology will determine the myriad of signals (mass-to-charge ratios) present in urine samples, which correspond to metabolites that become bioavailable after the intake of the test foods, collected at 0-1, 1-2, 4-6, 6-12, and 12-24 hours after intake. The analysis of the patterns in the metabolome will facilitate the discovery of potential biomarkers of intake.
Metabolic profiling of serum samples after intake of mango, amaranth, nopal, corn tortilla, avocado, and guava, detected as mass-to-charge signals (cps) by an untargeted metabolomics approach over 24 hours post-intake. | Before intake of foods 00 hours to 24 hours after intake.
  Given the absence of a priori knowledge of specific serum biomarkers of intake for mango, nopal, amaranth, avocado, corn tortilla, and guava, an untargeted metabolomics approach will be employed to identify them. As an exploratory approach, this methodology will determine the myriad of signals (mass-to-charge ratios) present in serum samples collected at baseline, 1 hour, 2 hours, 4 hours, 6 hours, and 24 hours after the intake of. The analysis of the patterns in the metabolome will facilitate the discovery of potential biomarkers of intake.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Vázquez Manjarrez, PhD, Principal Investigator — National Institute of Medical Sciences and Nutrition Salvador Zubirán
Locations (1):
- Instituto de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

REFERENCES:
- [Background] Archer E, Marlow ML, Lavie CJ. Controversy and debate: Memory-Based Methods Paper 1: the fatal flaws of food frequency questionnaires and other memory-based dietary assessment methods. J Clin Epidemiol. 2018 Dec;104:113-124. doi: 10.1016/j.jclinepi.2018.08.003. Epub 2018 Aug 17. PMID 30121379
- [Background] Tinker LF, Sarto GE, Howard BV, Huang Y, Neuhouser ML, Mossavar-Rahmani Y, Beasley JM, Margolis KL, Eaton CB, Phillips LS, Prentice RL. Biomarker-calibrated dietary energy and protein intake associations with diabetes risk among postmenopausal women from the Women's Health Initiative. Am J Clin Nutr. 2011 Dec;94(6):1600-6. doi: 10.3945/ajcn.111.018648. Epub 2011 Nov 9. PMID 22071707
- [Background] Vanderslice JT, Higgs DJ. Vitamin C content of foods: sample variability. Am J Clin Nutr. 1991 Dec;54(6 Suppl):1323S-1327S. doi: 10.1093/ajcn/54.6.1323s. PMID 1962591
- [Background] Andersen MB, Kristensen M, Manach C, Pujos-Guillot E, Poulsen SK, Larsen TM, Astrup A, Dragsted L. Discovery and validation of urinary exposure markers for different plant foods by untargeted metabolomics. Anal Bioanal Chem. 2014 Mar;406(7):1829-44. doi: 10.1007/s00216-013-7498-5. Epub 2014 Jan 4. PMID 24390407
- [Background] Gibbons H, Michielsen CJR, Rundle M, Frost G, McNulty BA, Nugent AP, Walton J, Flynn A, Gibney MJ, Brennan L. Demonstration of the utility of biomarkers for dietary intake assessment; proline betaine as an example. Mol Nutr Food Res. 2017 Oct;61(10). doi: 10.1002/mnfr.201700037. Epub 2017 Jul 20. PMID 28556565
- [Background] Cuparencu C, Rinnan A, Dragsted LO. Combined Markers to Assess Meat Intake-Human Metabolomic Studies of Discovery and Validation. Mol Nutr Food Res. 2019 Sep;63(17):e1900106. doi: 10.1002/mnfr.201900106. Epub 2019 Jun 13. PMID 31141834
- [Background] Vazquez-Manjarrez N, Weinert CH, Ulaszewska MM, Mack CI, Micheau P, Petera M, Durand S, Pujos-Guillot E, Egert B, Mattivi F, Bub A, Dragsted LO, Kulling SE, Manach C. Discovery and Validation of Banana Intake Biomarkers Using Untargeted Metabolomics in Human Intervention and Cross-sectional Studies. J Nutr. 2019 Oct 1;149(10):1701-1713. doi: 10.1093/jn/nxz125. PMID 31240312
- [Background] Giesbertz P, Brandl B, Lee YM, Hauner H, Daniel H, Skurk T. Specificity, Dose Dependency, and Kinetics of Markers of Chicken and Beef Intake Using Targeted Quantitative LC-MS/MS: A Human Intervention Trial. Mol Nutr Food Res. 2020 Mar;64(5):e1900921. doi: 10.1002/mnfr.201900921. Epub 2020 Jan 29. PMID 31916678
- [Background] Ulaszewska MM, Weinert CH, Trimigno A, Portmann R, Andres Lacueva C, Badertscher R, Brennan L, Brunius C, Bub A, Capozzi F, Cialie Rosso M, Cordero CE, Daniel H, Durand S, Egert B, Ferrario PG, Feskens EJM, Franceschi P, Garcia-Aloy M, Giacomoni F, Giesbertz P, Gonzalez-Dominguez R, Hanhineva K, Hemeryck LY, Kopka J, Kulling SE, Llorach R, Manach C, Mattivi F, Migne C, Munger LH, Ott B, Picone G, Pimentel G, Pujos-Guillot E, Riccadonna S, Rist MJ, Rombouts C, Rubert J, Skurk T, Sri Harsha PSC, Van Meulebroek L, Vanhaecke L, Vazquez-Fresno R, Wishart D, Vergeres G. Nutrimetabolomics: An Integrative Action for Metabolomic Analyses in Human Nutritional Studies. Mol Nutr Food Res. 2019 Jan;63(1):e1800384. doi: 10.1002/mnfr.201800384. Epub 2018 Oct 11. PMID 30176196
- [Background] Dragsted LO, Gao Q, Scalbert A, Vergeres G, Kolehmainen M, Manach C, Brennan L, Afman LA, Wishart DS, Andres Lacueva C, Garcia-Aloy M, Verhagen H, Feskens EJM, Pratico G. Validation of biomarkers of food intake-critical assessment of candidate biomarkers. Genes Nutr. 2018 May 30;13:14. doi: 10.1186/s12263-018-0603-9. eCollection 2018. PMID 29861790
- [Background] Barnes RC, Krenek KA, Meibohm B, Mertens-Talcott SU, Talcott ST. Urinary metabolites from mango (Mangifera indica L. cv. Keitt) galloyl derivatives and in vitro hydrolysis of gallotannins in physiological conditions. Mol Nutr Food Res. 2016 Mar;60(3):542-50. doi: 10.1002/mnfr.201500706. Epub 2016 Feb 2. PMID 26640139
- [Background] Kim H, Castellon-Chicas MJ, Arbizu S, Talcott ST, Drury NL, Smith S, Mertens-Talcott SU. Mango (Mangifera indica L.) Polyphenols: Anti-Inflammatory Intestinal Microbial Health Benefits, and Associated Mechanisms of Actions. Molecules. 2021 May 6;26(9):2732. doi: 10.3390/molecules26092732. PMID 34066494
- [Background] Ferreira CM, Vieira AT, Vinolo MA, Oliveira FA, Curi R, Martins Fdos S. The central role of the gut microbiota in chronic inflammatory diseases. J Immunol Res. 2014;2014:689492. doi: 10.1155/2014/689492. Epub 2014 Sep 18. PMID 25309932
- [Background] Dreher ML, Davenport AJ. Hass avocado composition and potential health effects. Crit Rev Food Sci Nutr. 2013;53(7):738-50. doi: 10.1080/10408398.2011.556759. PMID 23638933
- [Background] Fulgoni VL 3rd, Dreher M, Davenport AJ. Avocado consumption is associated with better diet quality and nutrient intake, and lower metabolic syndrome risk in US adults: results from the National Health and Nutrition Examination Survey (NHANES) 2001-2008. Nutr J. 2013 Jan 2;12:1. doi: 10.1186/1475-2891-12-1. PMID 23282226
- [Background] Vazquez-Manjarrez N, Ulaszewska M, Garcia-Aloy M, Mattivi F, Pratico G, Dragsted LO, Manach C. Biomarkers of intake for tropical fruits. Genes Nutr. 2020 Jun 19;15(1):11. doi: 10.1186/s12263-020-00670-4. PMID 32560627
- [Background] Qin XJ, Yu Q, Yan H, Khan A, Feng MY, Li PP, Hao XJ, An LK, Liu HY. Meroterpenoids with Antitumor Activities from Guava (Psidium guajava). J Agric Food Chem. 2017 Jun 21;65(24):4993-4999. doi: 10.1021/acs.jafc.7b01762. Epub 2017 Jun 9. PMID 28578580
- [Background] Kohlert C, van Rensen I, Marz R, Schindler G, Graefe EU, Veit M. Bioavailability and pharmacokinetics of natural volatile terpenes in animals and humans. Planta Med. 2000 Aug;66(6):495-505. doi: 10.1055/s-2000-8616. PMID 10985073
- [Background] Pujos-Guillot E, Hubert J, Martin JF, Lyan B, Quintana M, Claude S, Chabanas B, Rothwell JA, Bennetau-Pelissero C, Scalbert A, Comte B, Hercberg S, Morand C, Galan P, Manach C. Mass spectrometry-based metabolomics for the discovery of biomarkers of fruit and vegetable intake: citrus fruit as a case study. J Proteome Res. 2013 Apr 5;12(4):1645-59. doi: 10.1021/pr300997c. Epub 2013 Mar 5. PMID 23425595
- [Background] Lopez-Romero P, Pichardo-Ontiveros E, Avila-Nava A, Vazquez-Manjarrez N, Tovar AR, Pedraza-Chaverri J, Torres N. The effect of nopal (Opuntia ficus indica) on postprandial blood glucose, incretins, and antioxidant activity in Mexican patients with type 2 diabetes after consumption of two different composition breakfasts. J Acad Nutr Diet. 2014 Nov;114(11):1811-8. doi: 10.1016/j.jand.2014.06.352. Epub 2014 Aug 12. PMID 25132122
- [Background] Vazquez-Manjarrez N, Guevara-Cruz M, Flores-Lopez A, Pichardo-Ontiveros E, Tovar AR, Torres N. Effect of a dietary intervention with functional foods on LDL-C concentrations and lipoprotein subclasses in overweight subjects with hypercholesterolemia: Results of a controlled trial. Clin Nutr. 2021 May;40(5):2527-2534. doi: 10.1016/j.clnu.2021.02.048. Epub 2021 Mar 6. PMID 33932799
- [Background] Nkobole N, Prinsloo G. 1H-NMR and LC-MS Based Metabolomics Analysis of Wild and Cultivated Amaranthus spp. Molecules. 2021 Feb 4;26(4):795. doi: 10.3390/molecules26040795. PMID 33557008
- [Background] Warrack BM, Hnatyshyn S, Ott KH, Reily MD, Sanders M, Zhang H, Drexler DM. Normalization strategies for metabonomic analysis of urine samples. J Chromatogr B Analyt Technol Biomed Life Sci. 2009 Feb 15;877(5-6):547-52. doi: 10.1016/j.jchromb.2009.01.007. Epub 2009 Jan 14. PMID 19185549
- [Background] Kohl SM, Klein MS, Hochrein J, Oefner PJ, Spang R, Gronwald W. State-of-the art data normalization methods improve NMR-based metabolomic analysis. Metabolomics. 2012 Jun;8(Suppl 1):146-160. doi: 10.1007/s11306-011-0350-z. Epub 2011 Aug 12. PMID 22593726
- [Background] Scalbert A, Brennan L, Manach C, Andres-Lacueva C, Dragsted LO, Draper J, Rappaport SM, van der Hooft JJ, Wishart DS. The food metabolome: a window over dietary exposure. Am J Clin Nutr. 2014 Jun;99(6):1286-308. doi: 10.3945/ajcn.113.076133. Epub 2014 Apr 23. PMID 24760973
- [Background] van den Berg RA, Hoefsloot HC, Westerhuis JA, Smilde AK, van der Werf MJ. Centering, scaling, and transformations: improving the biological information content of metabolomics data. BMC Genomics. 2006 Jun 8;7:142. doi: 10.1186/1471-2164-7-142. PMID 16762068
- [Background] Vinaixa M, Samino S, Saez I, Duran J, Guinovart JJ, Yanes O. A Guideline to Univariate Statistical Analysis for LC/MS-Based Untargeted Metabolomics-Derived Data. Metabolites. 2012 Oct 18;2(4):775-95. doi: 10.3390/metabo2040775. PMID 24957762
- See also: The Food database — http://foodb.ca/